CLINICAL TRIAL: NCT06396806
Title: A Prospective, Randomized, Open, Parallel-controlled, Superior-efficacy Clinical Study of Radical Sigmoidectomy for Sigmoid Cancer Versus Radical Sigmoidectomy Combined with Indocyanine Green Fluorescence Imaging Lymphatic Tracing Dissection in the Treatment of Sigmoid Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Chief physician，Assistant to the dean, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-35
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Sigmoid Cancer
MeSH Terms: conditions — Sigmoid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- radical sigmoidectomy (No Intervention): radical sigmoidectomy
- radical sigmoidectomy combined with indocyanine green fluorescence imaging (Experimental): At the end of routine operation, indocyanine green was used for lymph node tracing, and further lymph node dissection was performed according to the tracer results.
  Interventions: Procedure: indocyanine green fluorescence imaging lymphatic tracing

INTERVENTIONS:
Procedure: indocyanine green fluorescence imaging lymphatic tracing — At the end of routine operation, indocyanine green was used for lymph node tracing, and further lymph node dissection was performed according to the tracer results.
  Arms: radical sigmoidectomy combined with indocyanine green fluorescence imaging

SUMMARY:
he purpose of this study is to explore the clinical outcomes of Indocyanine Green Tracer using in laparoscopic radical sigmoidectomy for sigmoid adenocarcinoma (cT2-T4a N0 M0，T1-T4a N+ M0).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old
2. Confirmed sigmoid adenocarcinoma cancer pathologically
3. Location of tumor: the sigmoid colon (descending colon from vertical to horizontal point) is the starting point of sigmoid colon, and the end point of sigmoid colon is at 15cm of anal margin.
4. CT showed sigmoid colon cancer: T3-4a N+ M0
5. Patients with non-local recurrence or distant metastasis;
6. no multiple colorectal cancer;
7. no neoadjuvant therapy;
8. physical conditions such as heart, lung, liver and kidney function can tolerate surgery.
9. Willing and able to provide written informed consent for participation in this study

Exclusion Criteria:

1. Complicated with other malignant tumors or previous history of malignant tumors;
2. patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc.;
3. patients with tumor invasion or involvement of adjacent organs requiring combined organ resection;
4. patients with poor anal function and incontinence before operation;
5. patients with inflammatory bowel disease or familial adenomatous polyposis
6. ASA grade ≥ IV and / or ECOG physical status score > 2;
7. patients with severe hepatorenal function, cardiopulmonary function, blood coagulation dysfunction or severe underlying diseases unable to tolerate surgery;
8. history of severe mental illness;
9. pregnant or lactating women;
10. patients with uncontrolled infection before operation;
11. patients with other clinical and laboratory conditions considered by some researchers should not participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate | 3 years after the surgery
  odisease-free survival was defined as the time from surgery to the time of recurrence or death from any cause

SECONDARY OUTCOMES:
Total number of retrieved lymph nodes | 14 days after the surgery
  Compare total number of retrieved lymph nodes in both group
Number of Metastasis Lymph Nodes | 14 days after the surgery
  Compare number of positive lymph nodes in both group.
The number of lymph nodes at each station | 14 days after the surgery
The rate of fluorescence | 14 days after the surgery
  The number of fluorescent lymph node in experimental group is divided by the total number of lymph nodes in active experimental group
Positive rate | 14 days after the surgery
  The number of positive lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes in experimental group
False positive rate | 14 days after the surgery
  The number of negative lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes in experimental group
Negative rate | 14 days after the surgery
  The number of negative lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes in experimental group
False negative rate | 14 days after the surgery
  The number of positive lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes in experimental group
Morbidity rate | 30 days after the surgery
  This is for the early postoperative complication
mortality rate | 30 days after the surgery
  mortality, which defined as the event observed within 30 days after surgery
Pathological outcomes checklist | 14 days after the surgery
  Quality of the mesorectum specimen, number of harvested lymph nodes, status of circumferential resection margin, and distal resection margin
3-year Overall survival rate | 3 years after the surgery
  Overall survival was defined as the time from surgery to death from any cause
5-year Overall survival rate | 5 years after the surgery
  Overall survival was defined as the time from surgery to death from any cause
5-year Disease-free survival rate | 5 years after the surgery
Local recurrence rate | 3 years after the surgery
  Local recurrence was defined as radiologic or histopathologic evidence of any recurrent disease deposit located in the pelvis in the prior area of dissection following a primary rectal cancer resection, with or without distal metastasis.
Postoperative function (voiding function, sexual function) and quality of life | 3 years after the surgery
The correlation between the number of lymph nodes and 3-year overall survival rate and 3-year disease-free survival rate | 3 years after the surgery
Minimal Residual Disease, MRD | 3 years after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University, Sixth Affiliated Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided